CLINICAL TRIAL: NCT01299311
Title: The Effect of Activity on Insulin Sensitivity and Lipid Metabolism in Sedentary, Overweight People.
Brief Title: NEAT and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MEC 10-2-057
Record Dates: First submitted 2011-01-17; First posted 2011-02-18 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Overweight
Keywords: insulin sensitivity
MeSH Terms: conditions — Overweight; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Inactivity (No Intervention): 4 days of inactivity, mainly sitting
- NEAT (Active Comparator): 4 days of NEAT (everyday activities)
  Interventions: Behavioral: NEAT
- Exercise (Active Comparator): 4 days of inactivity combined with 1 hour of exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: NEAT — 4 days of everyday activities, including 4 hours of walking, 8 hours of sitting, 2 hours of standing, 2 hours of everyday activities and 8 hours of sleeping or laying down per day
  Arms: NEAT
Behavioral: Exercise — 4 days of activity program, including 1 hour biking (exercise), 13 hours of sitting, 2 hours of everyday activities and 8 hours of sleeping or laying down per day
  Arms: Exercise

SUMMARY:
The effect of Non-Exercise Activity Thermogenesis (NEAT) or inactivity on insulin sensitivity and lipid metabolism is unclear. Research recently published shows that activities associated with everyday activities, summarized as NEAT, such as walking and standing, have a much greater role in energy expenditure than exercise. Therefore, the objective of the present study is to evaluate the effect of 4 days of inactivity (mainly sitting), 4 days of everyday activities (sitting, walking and standing), and 4 days of inactivity and exercise (sitting and biking) on glucose metabolism and insulin sensitivity using an oral glucose tolerance test, and on lipid metabolism in sedentary, overweight people. The investigators hypothesize that:

1. 4 days of everyday activities (NEAT) will cause an increased glucose tolerance and increased insulin sensitivity compared to 4 days of inactivity in sedentary, overweight people.
2. 4 days of exercise will improve glucose tolerance and insulin sensitivity more than 4 days of NEAT with equal energy expenditure, in sedentary, overweight people.
3. Fasting triglyceride will have the same course as glucose, mentioned in 1. and 2.

DETAILED DESCRIPTION:
To evaluate the effect of Non-Exercise Activity Thermogenesis (NEAT) on glucose and lipid metabolism in sedentary, overweight people, the subjects included in the study protocol will follow 3 times a certain activity program of 4 days. These activity programs are:

* Inactivity: 14 hours of sitting, 2 hours of everyday activities, 8 hours of sleeping or laying down per day.
* NEAT: 4 hours of walking, 8 hours of sitting, 2 hours of standing, 2 hours of everyday activities, 8 hours of sleeping or laying down per day.
* Exercise: 1 hour biking, 13 hours of sitting, 2 hours of everyday activities, 8 hours of sleeping or laying down per day.

The subjects will be biking using a home trainer, measuring energy expenditure, and supervised by one of the members of the research team. They will bike until they have reached a certain amount of kCal. The subjects will wear two accelerometers during all 3 activity programs to evaluate the amount of each activity (sitting, walking, standing, laying/sleeping). The Computer Science and Applications (CSA) Actigraph accelerometer will be placed on the back and the Continuous Activity Monitor (CAM) Maastricht instrument on the leg. Furthermore, the subjects will be requested to note their activities and dietary intake in a diary. After every 4 days of each activity program, an oral glucose tolerance test will be performed in the morning (fasting state) of the next day (day 5). Before and 15, 30, 45, 60, 90, 120 minutes after ingestion of 75 gram of glucose in water, blood will be drawn for measurements of glucose and insulin. Only at baseline (t=0 minutes), blood will be drawn to measure cholesterol, HDL, LDL, triglycerides, apoA and apoB.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-30 years old
* BMI between 25.0-30.0 kg/m2
* Sedentary, defined as maximum of exercise of 1 hour/week and less than 2x/week

Exclusion Criteria:

* Cardiovascular disease
* Diabetes mellitus type 1 or 2 or fasting glucose > 6.9 mmol/L
* Other diseases that make physical activity difficult
* Alcohol > 2 consumptions/day
* Illegal drug use and cannabis use
* Medication use, other than contraception
* Triglycerides > 3.0 mmol/L

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity after 4 days of NEAT compared to 4 days of inactivity and compared to 4 days of exercise | day 5
  Change in insulin sensitivity measured using oral glucose tolerance test

SECONDARY OUTCOMES:
Change in fasting triglycerides after 4 days of NEAT compared to 4 days of inactivity and compared to 4 days of exercise | 5 day

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas C Schaper, Prof., MD, Principal Investigator — Maastricht University Medical Center/ University of Maastricht
Locations (1):
- Maastricht University Medical Center/ University of Maastricht, Maastricht, Netherlands